CLINICAL TRIAL: NCT05549336
Title: Single-center, Prospective Cohort Study of PD-1inhibitors on Clinical Outcomes of Carotid Plaques in Tumor Patients
Brief Title: Single-center, Prospective Cohort Study of PD-1 Inhibitors on Clinical Outcomes of Carotid Plaques in Tumor Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0803
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Carotid Artery Plaque; Pd-1 Inhibitors
MeSH Terms: conditions — Carotid Stenosis | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD-1-treated tumor patients: Tumor patients who are initiating receive chemotherapy that includes PD-1 inhibitors.
  Interventions: Drug: PD-1 inhibitor
- non-PD-1-treated tumor patients: Tumor patients who are initiating receive chemotherapy that not includes PD-1 inhibitors.

INTERVENTIONS:
Drug: PD-1 inhibitor — PD-1 inhibitor is defined as the exposure factor in our cohort study, for the tumor patients with the treatment of PD-1 inhibitor are allocated to the Exposure group whereas those tumor patients without the treatment of PD-1 inhibitor are allocated to the Non-exposure group.
  Other Names: PD-1 immune checkpoint blockades
  Groups: PD-1-treated tumor patients

SUMMARY:
This is a single-center, prospective cohort study on the comparison of clinical outcomes of carotid plaques in PD-1-treated tumor patients vs non-PD-1-treated tumor patients.

DETAILED DESCRIPTION:
Atherosclerosis, a chronic inflammatory disorder, leads to cardio-cerebrovascular diseases, causing most of the global deaths. The chronic and non-resolved inflammatory responses of both innate and adaptive immune cells are involved in the all-stage pathogenesis of atherosclerosis. The impairment of inflammatory resolution promotes atherogenesis and causes instability of atherosclerotic plaques. Their subsequent rupture would induce severe cardio-cerebrovascular incidences (e.g., acute myocardial infarction and ischemic strokes). Recent progress in anti-inflammatory immunotherapies on human atherosclerosis opens the door to resolving this inflammatory disorder by targeting the immune system. However, the impacts of PD-1 immune checkpoint blockades on the progressions of human carotid plaques are not determined yet.

This is a prospective cohort study, which aims to evaluate the effectiveness of PD-1 immune checkpoint blockades on atherosclerotic carotid plaques in tumor patients in comparison to those with non-PD-1-treated tumor patients. The method for quantification and evaluation of atherosclerotic plaques are based on: (1) the mean intima-media thickness of the common carotid artery (Mean CCA thickness); (2) the maximum intima-media thickness of the internal carotid artery (maximum ICA thickness); (3) Carotid plaque areas: by calculation of the plaque area of atherosclerotic plaques on the long axis direction of artery on the ultrasound images. By comparing the above-mentioned parameters at the same location of the carotid artery in the patients when initiating the first dose of anti-PD-1 or non-PD-1 chemotherapy and 3 months after anti-PD-1 or non-PD-1 chemotherapy. It is designed to assess the effectiveness of PD-1 immune checkpoint blockades or non-PD-1 chemotherapy on the clinical prognosis of carotid plaques after a period of 3-month treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects know about the experiment and signed the informed consent voluntarily; and
2. Subjects are tumor patients and all kinds of tumor diseases of subjects are acceptable; and
3. Subjects are initiating to receive chemotherapy; and
4. Subjects are diagnosed with atherosclerotic carotid plaques by ultrasound examination at the timepoint of the first-dose treatment; and

Exclusion Criteria:

1. Subjects stop receiving or changing the existing chemotherapy during follow-up; or
2. Subjects are reluctant to continue to be involved in this study; or
3. Subjects are known pregnant and lactating women; or
4. Subjects are not complicated with atherosclerotic carotid plaques at the timepoint of the first-dose treatment; or

4. The parameters (e.g., CCA intima-media, ICA intima-media, or carotid plaque area) could not be calculated because of the quality of the ultrasound image; or 5. Other situations that the researchers judged are not suitable for further inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All tumor patients who are initiating the chemotherapy in The Second Affiliated Hospital, Zhejiang University School of Medicine (SAHZU) and willing to join this cohort study after the date of recruiting (19th Sep 2022). These patients who are eligible for the inclusion criteria would be the targets for further follow-up.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Carotid plaque area | 3 months
  Carotid plaque area measured by ultrasound (cross-sectional area of longitudinal views of all plaques seen) to quantify the increase or decrease of atherosclerotic carotid plaques.
The mean intima-media thickness of the common carotid artery | 3 months
  It was measured over a segment of the common carotid artery that was 1 cm long, located approximately 0.5 cm below the carotid-artery bulb, and considered not to contain any plaque (i.e., not to have any perceivable protrusion of the artery wall into the lumen).
The maximum intima-media thickness of the internal carotid artery | 3 months
  It was defined as the greatest intima-media thickness in either the right or left internal carotid artery extending from the bulb to 1 cm above the carotid sinus, ascertained from a total of four views on each side.

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD, PhD, Study Chair — 2nd Affiliated Hospital, School of Medicine at Zhejiang University; Lin Fan, PhD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine at Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spence JD, Eliasziw M, DiCicco M, Hackam DG, Galil R, Lohmann T. Carotid plaque area: a tool for targeting and evaluating vascular preventive therapy. Stroke. 2002 Dec;33(12):2916-22. doi: 10.1161/01.str.0000042207.16156.b9. PMID 12468791
- [Background] Lorenz MW, Polak JF, Kavousi M, Mathiesen EB, Volzke H, Tuomainen TP, Sander D, Plichart M, Catapano AL, Robertson CM, Kiechl S, Rundek T, Desvarieux M, Lind L, Schmid C, DasMahapatra P, Gao L, Ziegelbauer K, Bots ML, Thompson SG; PROG-IMT Study Group. Carotid intima-media thickness progression to predict cardiovascular events in the general population (the PROG-IMT collaborative project): a meta-analysis of individual participant data. Lancet. 2012 Jun 2;379(9831):2053-62. doi: 10.1016/S0140-6736(12)60441-3. Epub 2012 Apr 27. PMID 22541275
- [Background] Spence JD. Measurement of carotid plaque burden. JAMA Neurol. 2015 Apr;72(4):383-4. doi: 10.1001/jamaneurol.2014.3002. No abstract available. PMID 25686472
- [Background] Lechareas S, Yanni AE, Golemati S, Chatziioannou A, Perrea D. Ultrasound and Biochemical Diagnostic Tools for the Characterization of Vulnerable Carotid Atherosclerotic Plaque. Ultrasound Med Biol. 2016 Jan;42(1):31-43. doi: 10.1016/j.ultrasmedbio.2015.09.003. Epub 2015 Oct 20. PMID 26493239
- [Background] Polak JF, Pencina MJ, Pencina KM, O'Donnell CJ, Wolf PA, D'Agostino RB Sr. Carotid-wall intima-media thickness and cardiovascular events. N Engl J Med. 2011 Jul 21;365(3):213-21. doi: 10.1056/NEJMoa1012592. PMID 21774709